CLINICAL TRIAL: NCT02947997
Title: Pilot Study for Imaging of the Esophagus Using Tethered Capsule OCT Endomicroscopy With Distal Scanning
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2015-P000777
Record Dates: First submitted 2016-04-14; First posted 2016-10-28 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- OFDI capsule imaging: Subject will swallow the OFDI capsule and imaging will be acquired using the OFDI imaging system.
  Interventions: Device: OFDI capsule

INTERVENTIONS:
Device: OFDI capsule — Imaging of esophagus using OFDI capsule and system

SUMMARY:
The purpose of this study is to test feasibility of a redesigned tethered capsule catheter that contains an integrated micro-motor. Investigators will be testing imaging of this new technology in healthy volunteers.

DETAILED DESCRIPTION:
10 healthy volunteers will be enrolled and asked to swallow the Distal Scanning Capsule. The subjects will be awake and un-sedated.

The capsule is attached to a string like tether which allows the operator to control as well as navigate the capsule as it progresses down the esophagus using natural propulsive force called peristalsis.

As the capsule progresses through the esophagus, multiple images of the esophagus are acquired in real time to be analyzed later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be over the age of 18
* Subjects must be able to give informed consent
* Subjects must have no solid food for 4 hours prior to the procedure, and only clear liquids for 2 hours prior to the procedure.

Exclusion Criteria:

* Subjects with the inability to swallow pills and capsules.
* Esophageal fistula and/or esophageal strictures with a stricture diameter that is smaller than the diameter of the capsule.
* Subjects who have a bleeding disorder and are currently on anti-coagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events occurred after participants enrollment.
Period: Overall Study
Arm/Group | OFDI Capsule Imaging
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OFDI Capsule Imaging
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (5.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants For Whom Good Quality Images Were Recorded After Swallowing The OFDI Capsule
Description: An investigator to assess the quality of the recorded images obtained with each exam after imaging has been completed
Time Frame: Approximate 20 minute visit (5 min image acquisition)
Measure: Count of Participants; unit: Participants
Groups:
- OFDI Capsule Imaging: Subjects who swallowed the OFDI capsule and good quality imaging was acquired using the OFDI imaging system.
Arm/Group | OFDI Capsule Imaging
Number analyzed (Participants) | 4
Participants | 3

ADVERSE EVENTS:
Arm/Group | OFDI Capsule Imaging
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No